CLINICAL TRIAL: NCT00218933
Title: Anti-remodeling Effect of High-intensity Interval Training in Patients With Post-infarction Heart Failure on Optimal Treatment
Brief Title: High-intensity Exercise Training in Patients With Post-infarction Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HFEX-1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: Interval training; Endothelial dysfunction; Aerobic capacity; Exercise
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- moderate exercise training (Active Comparator)
  Interventions: Behavioral: Moderate intensity exercise training
- high intensity exercise training (Experimental)
  Interventions: Behavioral: High intensity exercise training
- controls (No Intervention)

INTERVENTIONS:
Behavioral: Moderate intensity exercise training — 12-weeks, 2-3 times per week moderate exercise-intensity (70% of peak heart rate)
  Arms: moderate exercise training
Behavioral: High intensity exercise training — 12-weeks, 2-3 times per week high-intensity interval-training (95% of peak heart rate)
  Arms: high intensity exercise training

SUMMARY:
Introduction: Moderate-intensity endurance-training is known to reduce symptoms, increase exercise tolerance, and improve quality of life in patients with chronic heart failure. The training benefits have mainly been attributed to adaptations in the peripheral circulation and skeletal muscle rather than to adaptations in cardiac performance. However attenuation of left ventricular (LV) remodelling has been documented in some studies. The effects of high- vs. moderate exercise-intensity on LV-remodelling and endothelial function in patients with post-infarction heart failure are not definitively established and were studied in the present study.

Methods: Patients with post-infarction heart failure (45-87 yrs, 22-males, 5-females, all received b-blockers and ACE-inhibitors, EF 29%, peak oxygen uptake 13 ml/kg/min) were randomized to 12-weeks, 2-3 times per week, of either moderate exercise-intensity (70% of peak heart rate), high-intensity interval-training (95% of peak heart rate) or to a control group that received advise from their regular doctors. Patients in the two exercise-groups covered similar distance on the treadmill at each exercise-session so that only exercise-intensity differed; i.e. the duration of exercise was longer in the moderate-intensity group. Ultrasound was used to assess LV-dimension and function (including Tissue Doppler Imaging, TDI) and endothelial function in the brachial-artery.

ELIGIBILITY:
Inclusion Criteria:

Post-infarction heart failure and optimal treatment (ACE-inhibitors, Beta-blockade)

Exclusion Criteria:

Not able to walk on a treadmill, unstable angina, participating in another experiment, serious arrhythmia

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-10 (Actual); Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Remodelling of heart function and structure | 3 months

SECONDARY OUTCOMES:
Improved endothelial and skeletal muscle as well as quality of life | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisloff, Ph.D, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726